CLINICAL TRIAL: NCT00475631
Title: Economic Evaluation of Clubfoot Treatment: One Centre's Experience
Status: Withdrawn | Type: Observational
Why Stopped: The person who started the study joined medical school
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christine Alvarez, Principle Investigator, University of British Columbia
Other Study IDs: H03-70532
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2017-05

CONDITIONS: Clubfoot
Keywords: Clubfoot; Chart review
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose:

The purpose of the study is to complete a cost analysis of the different methods used for clubfoot treatment.

Objectives:

Short-term objective: To explore the experience of British Columbia Children's Hospital (BCCH) with costs and outcomes related to the various forms of clubfoot management since 1984 to present.

Long-term objective: To use the information gathered in this project and apply it to future studies in the clubfoot research program and to do a complete cost-benefit analysis.

Hypothesis: The hypothesis of the study is that the BCCH clubfoot treatment program has better outcomes in terms of reduced financial costs than the traditional surgical management.

DETAILED DESCRIPTION:
Inclusion criteria:

All patients who were diagnosed and treated for idiopathic clubfoot at BCCH between January 1984 and present are eligible for the study. Patients whose clubfoot is a secondary diagnosis to another disorder (mal-position, neuromuscular disorder and chromosomal abnormality) are excluded from this study.

Database design:

Using information gathered from literature review and interviews with several of the orthopaedic surgeons at BCCH the most common treatment methods for clubfoot and the ones that are and have been in use in BCCH were identified. Six treatment methods were then described in detail. These treatment methods are: comprehensive release, posterio-medial release, posterior release, Kite-method, Ponseti-method and BCCH-method. From all different treatment-steps possible "units" were designed. The units that were designed are: initial consult, clinic visit, consult physiotherapist, consult occupational therapist, OT-splint, consult orthotist, X-ray, Boots and Bars, AFO by orthotist, custom orthotic, shoes, surgery, cast applied during surgery, surgery second foot, surgery extra, anaesthesia extra 1-3, daycare surgery, overnight stay in hospital, gastrosoleus defunctioning using Botox, Botox, gait analysis and non-clubfoot related hospital encounter. Per unit there are more treatment "options" available. For example in the unit "clinic visit", there are 18 options, such as clinic visit, clinic visit with manipulation and casting using plaster of paris below knee, clinic visit with manipulation and casting using plaster of paris above knee, clinic visit with manipulation and casting using 3-M soft cast below knee. Within the unit "X-ray" there are 3 options such as unilateral X-ray of the foot, bilateral X-ray of the foot, X-ray of the pelvis.

More units were designed that are not part of the treatment, but do have their impact on the costs concerning the treatment and therefore have to be considered. These units are: number of persons traveling, days away form home, lost wages, air transportation, ground transport, mileage, accommodation and meals.

All these units, together with patient demographics (patient ID, last name, first name, gender, hometown and distance to BCCH) and intervention type (one of the 6 treatment-regimes that the patient fits in) formed the database, which was set up in the Microsoft Excel program.

Patient Data collection:

All patients that are eligible for this study were identified using the hospital data retrieval system. The patient's hospital medical records will be collected and chart review will be performed. Patient data will be entered into the database, using one line for every visit (either as an inpatient or as an outpatient) to the hospital.

Costing Data collection:

Direct costs: A detailed breakdown of all "parts" constituting the units was performed. Costing information on all these parts was then obtained using a great variety of sources, including the MSP-billing book, personal communication with a pharmacy- representative and interviews with nursing representatives, an expert in the financial department and experts in the decision support department.

General overhead costs: The general overhead costs will be determined using information from the decision support services and from the Orthopaedic department.

Data analysis: It is a cost analysis between the different methods of orthopaedic treatment for clubfoot. Statistical analysis will be completed on all continuous variables. Statistical analysis will be completed using SAS Statistical Software (SAS Institute, Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with clubfoot

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients who were diagnosed and treated for idiopathic clubfoot at BCCH between January 1984 and present are eligible for the study. Patients whose clubfoot is a secondary diagnosis to another disorder (mal-position, neuromuscular disorder and chromosomal abnormality) are excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, MD, Principal Investigator — University of British Columbia